CLINICAL TRIAL: NCT05653674
Title: The Effect of Acceptance and Commitment Approach-Based Psychoeducation on Nursing Students' Psychological Distress, Psychological Flexibility, Mindfullness and Values: A Randomized Control Trial
Brief Title: The Effect of Acceptance and Commitment Approach-Based Psychoeducation on Nursing Students' Psychological Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Neslihan Partlak Günüşen, Professor, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 6596-GOA
Record Dates: First submitted 2022-11-22; First posted 2022-12-16 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Psychological Distress
Keywords: Psychological Distress; Mindfullness; Values; Acceptance and commitment approach; Psychological flexibility; Psychiatric Nursing

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Experimental): The experimental group will consist of 40 students in total, 4 groups of 10 students each, and the students will receive face-to-face psychoeducation for 6 weeks, each session for 60 minutes.
  Interventions: Behavioral: Acceptance and commitment approach-based psychoeducation
- Control (No Intervention): The control group will not receive any intervention during the application period and will be put on waitlist.

INTERVENTIONS:
Behavioral: Acceptance and commitment approach-based psychoeducation — The psychoeducation based on acceptance and commitment approach reducing psychological distress in nursing students; It has been prepared to increase psychological flexibility, mindfullness and level valuing. A potential approach that has been shown to be effective in reducing psychological distress is one of the third generation cognitive behavioral therapies; acceptance and commitment therapy. Acceptance and commitment-based approaches encourage participants to change their relationship with their thoughts and physical sensations through acceptance, mindfullness, and value-based action mechanisms.
  Arms: Experiment

SUMMARY:
The study is planned to be conducted in a randomized controlled experimental design in accordance with CONSORT. The study is planned to be carried out at X Nursing Faculty between November 2022 and February 2024. The randomization list will be hidden from the students, and the group to which each student will be included will be revealed after they are included in the study. In order to determine which group the nursing students to be included in the study will be in, the "Layered Block Randomization" method will be used and they will be assigned to the experimental and control groups according to the stress scores they get from the DASS-21 scale. Assignment of intervention and control groups to conceal randomization information to avoid study bias; It will be done by an expert who was not involved in the research. The experimental group will consist of 40 students in total, 4 groups of 10 students each, and the students will receive face-to-face psychoeducation for 6 weeks, each session for 60 minutes. The control group will not receive any intervention during the application period and will be put on waitlist. After the psychoeducation, as a post-test, one month, six months and one year later, follow-up measurements will be applied face-to-face and by telephone to the students who have completed the psychoeducation, and the scores will be compared with the control group. Among the sampling criteria; Being a nursing student, getting at least 8 points (mild and above) from the stress sub-dimension of the DASS-21 scale; Exclusion criteria from the sample included starting psychiatric treatment in the last three months, having previously participated in an acceptance and commitment or mindfullness-based program. In the research, descriptive information form will be filled from the students. The level of psychological distress will be measured with the Depression, Anxiety and Stress Scale Short Form (DASS-21). Psychological flexibility will be measured with the Acceptance and Action Questionnaire-II , mindfullness with the Mindfull Attention Awareness Scale and the level of valuing with the Valuing Questionnaire . Validity and reliability studies of the scales were carried out. Institutional permission was obtained from the faculty where the research was conducted.

DETAILED DESCRIPTION:
It is emphasized that nursing students experience high levels of stress (Köse et al., 2021; Ching et al., 2020). Since nursing students are exposed to different stressors during their education and their stress levels are high, it is important to examine their psychological distress (Reverté Villarloya et al., 2021; Serçe et al., 2021). In the literature, it is emphasized that there is a need for interventions including methods such as psychological flexibility and mindfullness in order to reduce psychological distress in nursing students and strengthen them against difficult experiences (Ching et al.,2020; Ten Hoeve et al.,2017;Günüşen 2017). A potential approach that has been shown to be effective in reducing psychological distress and gaining psychological flexibility is one of the third generation cognitive behavioral therapies; acceptance and commitment approach. The aim of the study is to examine the effect of psychoeducation based on acceptance and commitment approach applied to nursing students on psychological distress, psychological flexibility, mindfullness and values. The study is planned to be conducted in a randomized controlled experimental design in accordance with CONSORT. The study is planned to be carried out at X Nursing Faculty between November 2022 and February 2024. Firstly, the Depression, Anxiety and Stress Scale Short Form (DASS-21) will be applied to the students studying at the X Nursing Faculty, and students who get at least 8 points from the stress sub-dimension of the form will be invited to work by e-mail and telephone. G power statistical analysis program was used in the sample calculation required for the study, Type I error was 0.05, Type II error was 0.20 (power 0.80). In the analysis, it was determined that 25 students should be taken for each group. Considering that there may be losses, it is planned to include 80 students in total, 40 students in each group. The experimental group will consist of 40 students in total, 4 groups of 10 students each, and the students will receive face-to-face psychoeducation for 6 weeks, each session for 60 minutes. The control group will not receive any intervention during the application period and will be put on waitlist. After the completion of the research, if the initiative is determined to be effective, the program is planned to be applied to the volunteer students in the control group. After the psychoeducation, as a post-test, one month and six months late and one year, follow-up measurements will be applied face-to-face and by telephone to the students who have completed the psychoeducation, and the scores will be compared with the control group. The randomization list will be hidden from the students, and the group to which each student will be included will be revealed after they are included in the study. In order to determine which group the nursing students to be included in the study will be in, the "Layered Block Randomization" method will be used and they will be assigned to the experimental and control groups according to the stress scores they get from the DASS-21 scale. Assignment of intervention and control groups to conceal randomization information to avoid study bias; It will be done by an expert who was not involved in the research. Among the sampling criteria; Being a nursing student, getting at least 8 points (mild and above) from the stress sub-dimension of the DASS-21 scale; Exclusion criteria from the sample included starting psychiatric treatment in the last three months, having previously participated in an acceptance and commitment or mindfullness-based program. In the research, descriptive information form will be filled from the students. The level of psychological distress will be measured with the Depression, Anxiety and Stress Scale Short Form (DASS-21). Psychological flexibility will be measured with the Acceptance and Action Questionnaire-II , mindfullness with the Mindfull Attention Awareness Scale and the level of valuing with the Valuing Questionnaire . Validity and reliability studies of the scales were carried out. Institutional permission was obtained from the faculty where the research was conducted. The study was approved by the ethics committee of the relevant university (2021/26-08). The verbal and written consent will be obtained from the nursing students who will participate in the research; individuals will be informed that information about themselves will not be disclosed to others, and the "principle of confidentiality" will be followed. Nursing students will be informed about the purpose of the research and how to apply it. The primary researcher, who is not responsible for the education of the students, will lead the initiatives to protect the vulnerability of the students.There is no anticipated limitation of the study. The expenses of the study will be covered by the researcher. With this study, it is hoped that nursing students who participate in acceptance and commitment-based psychoeducation will participate in the health system in a more psychologically flexibility and strenghten way.

ELIGIBILITY:
Inclusion Criteria:

* Being a nursing student
* Getting at least 8 points (mild and above) from the stress sub-dimension of the DASS-21 scale

Exclusion Criteria:

-The sample included starting psychiatric treatment in the last three months Having previously participated in an acceptance and commitment or mindfullness-based program.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-02-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline psychological distress levels to the end point of the intervention and one month (4 weeks), six months (24 weeks), 12 months (48 weeks) after the intervention | Change from to the end point of the intervention and one month (4 weeks), six months (24 weeks), 12 months (48 weeks) after the intervention
  Depression, Anxiety and Stress Scale Short Form (DASS-21) the DASS-21 scale will be used to evaluate the psychological distress level of students. In this scale (DASS-21), there are seven questions each to measure the dimensions of depression, anxiety and stress. The first seven questions on the scale are about anxiety, seven questions between 8-14 are about depression and seven questions between 15-21 are about stress. The scale has a four-point Likert-type rating of 0 "not at all suitable for me", 1 "somewhat suitable for me", 2 "usually suitable for me", and 3 "completely suitable for me". While the lowest score that can be obtained for all dimensions in the scale is zero, the highest score can be 21.

SECONDARY OUTCOMES:
Change from baseline psychological flexibility levels to the end point of the intervention and one month (4 weeks), six months (24 weeks), 12 months (48 weeks) after the intervention | Change from to the end point of the intervention and one month (4 weeks), six months (24 weeks), 12 months (48 weeks) after the intervention
  Acceptance and Action Questionnaire-II (AAQ-II) The seven-item Acceptance and Action Questionnaire-II is a reliable and valid scale for measuring psychological flexibility in both clinical and non-clinical samples. The mean Cronbach Alpha coefficient was found to be .84, and the internal consistency was high.The questionnaire consists of seven items in total. The scale items are graded from 1 (never true) to 7 (always true). The lowest score to be taken from the scale is 7 and the highest score is 49. The AAQ-II is a seven-point Likert-type scale, and as the total score increases, psychological rigidity increases and psychological flexibility decreases
Change from baseline mindfullness levels to the end point of the intervention and one month (4 weeks), six months (24 weeks), 12 months (48 weeks) after the intervention | Change from to the end point of the intervention and one month (4 weeks), six months (24 weeks), 12 months (48 weeks) after the intervention
  Mindfull Attention Awareness Scale The Mindful Attention Awareness Scale was developed to measure the general level of mindfullness and attention to current processes in daily life. The Cronbach Alpha internal consistency coefficient calculated for the reliability of the scale is 0.80. The scale consists of 15 items. The lowest score that can be obtained from the scale is 15 and the highest 90. The scale is a 6-point Likert type scale: almost always (1), often (2), sometimes (3), rarely (4), rarely (5), almost never (6). The Mindful Attention Awareness Scale has a single factor and a single total score is obtained from the scale. As the score obtained from the scale increases, the level of mindfullness of the individual increases.
Change from baseline valuing levels to the end point of the intervention and one month (4 weeks), six months (24 weeks), 12 months (48 weeks) after the intervention | Change from to the end point of the intervention and one month (4 weeks), six months (24 weeks), 12 months (48 weeks) after the intervention
  The Valuing Questionnaire measures the extent to which people live in accordance with the value they have determined in the last week. The questionnaire is a Likert-type questionnaire consisting of 10 items and two sub-dimensions, "progression" and "obstruction". Progress sub-dimension emphasized being able to do daily tasks in line with values, while blocking sub-dimension emphasized living a life away from values in activities carried out for a week, unlike progress. The Cronbach's alpha value for the whole scale is 0.78. The lowest total score is zero, while the highest is 60. A high score indicates that individuals live a life in line with their values.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğçe Şık, Msc, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hayes SC. Acceptance and Commitment Therapy, Relational Frame Theory, and the Third Wave of Behavioral and Cognitive Therapies - Republished Article. Behav Ther. 2016 Nov;47(6):869-885. doi: 10.1016/j.beth.2016.11.006. Epub 2016 Nov 10. PMID 27993338